CLINICAL TRIAL: NCT03060187
Title: The "KU Score": Proposal and Clinical Evaluation of a Comprehensive Airway Exam Score; an Observational Study
Brief Title: Proposal and Clinical Evaluation of a Comprehensive Airway Exam Score
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12093
Record Dates: First submitted 2017-01-27; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Intubation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- KU Score: Participants asked to answer questions for the KU Score exam
  Interventions: Other: KU Score

INTERVENTIONS:
Other: KU Score — Exam with a max score of 10 and min score of 0. Designed as a preoperative assessment of the patient's airway.

SUMMARY:
The purpose of this observational study is to evaluate the usefulness of Kansas University airway exam score ("KU score") in predicting difficulty of placement of a breathing tube into the windpipe.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-IV
* Patients scheduled for a surgical or any other diagnostic or therapeutic procedure that requires endotracheal intubation (ETI)

Exclusion Criteria:

* Patients scheduled for an emergent surgery
* Obstetric patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will include persons presenting to the University of Kansas Hospital to have surgery under standard general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Correlation between KU score and intubation difficulty scale (IDS) measure | Time between preoperative exam to after intubation, up to 3 hours
  The measure is assessed during the time period between the start of preoperative examination on the day of surgery and completion of a standard tracheal intubation in the operating room. Correlation measured using the Spearman correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Mirsad Dupanović, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States